CLINICAL TRIAL: NCT01520194
Title: The Psychosocial and Economic Burden of Genital Warts for Women Attending Six Reproductive Health Clinics in Brazil
Brief Title: The Psychosocial and Economic Burden of Genital Warts
Acronym: GWburden
Status: Completed | Type: Observational
Sponsor: BEMFAM-Bem Estar Familiar (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BEMFAM 421
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Female Genital Warts
Keywords: genital warts; HPV; psychosocial burden; economic burden; female genital warts
MeSH Terms: conditions — Condylomata Acuminata; Financial Stress | interventions — Medical Records

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- psychosocial burden: 122 women attending reproductive health clinics were interwied using HPV Impact Profile (HIP) and a socio-economic characteristics questionnaire.
  Interventions: Other: women attending reproductive health clinics
- economic burden: Medical records of 102 patients diagnosed with genital warts were reviewed in the six BEMFAM's participating reproductive health clinics
  Interventions: Other: medical records

INTERVENTIONS:
Other: women attending reproductive health clinics — women visiting BEMFAM´s clinics from January 2012 until Narch 2013 filled a self-administered questionnaire based on psychometric scale developes by Zhu TC et al
  Groups: psychosocial burden
Other: medical records — medical chart review of patients assisted January 2009 to December 2010
  Groups: economic burden

SUMMARY:
Considering the importance of HPV(human papilomavirus) and related diseases in Brazil, and the lack of studies about both the economic and the psychosocial burden of these diseases, BEMFAM, a Brazilian non-governmental organization that provides reproductive health services and technical support to local governments proposes a study to measure the psychosocial and economic burden of genital warts.

DETAILED DESCRIPTION:
Cervical cancer is a public health issue in Brazil. The Cancer National Institute estimates that cervical cancer will be the second most incident among women, with 18.430 new cases in 2010. Human papillomavirus (HPV) is related to cervical cancer and is also responsible for benign lesions, such as genital warts.The Brazilian Ministry of Health estimates the prevalence of genital warts to be 5,7% among pregnant women and 21,5% among women attending sexually transmitted infections treatment clinics.The study will measure the psychosocial burden of genital warts using HPV Impact Profile questionnaire and the economic burden of genital warts among women attending its six reproductive health clinics.

There are two study objectives:

1 - to measure the psychosocial burden of genital warts in women attending six reproductive health clinics in Brazil. 2- to measure the economic burden of genital warts treatment for women attending six reproductive health clinics in Brazil.

Hypothesis testing:

For objective 1, the experiment compare differences on psychosocial burden of Genital Warts among subgroups and therefore does not include any formal hypothesis testing about the psychosocial burden of the disease in agreement with the extant literature on the subject (Xingshu Zhu et al., 2009).

Objective 2 aims to measure differentials in the economic burden of the disease among subgroups with different type of genital warts (newly diagnosed, recurrent and resistant), site of the lesion, age, duration of treatment, number of medical visits, type and number of medical procedures. No formal hypothesis will be tested.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18 to 45 years, who had a Pap-smear in the preceding 90 days or were diagnosed with genital warts during physical examination.
* good health

Exclusion Criteria:

* women self reported HIV-positive
* women undergoing antiretro-viral treatment
* illiteracy
* pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Reproductive health clinics
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
psychosocial burden of genital warts | January 2012 until March 2013
  122 individuals filled the self-administered questionnaire. Women with normal Pap smear presented lower scores of worries and concerns about gynecological health than women with cervical intraepithelial neoplasia or genital warts and higher scores of satisfaction with sexual life. Feelings of anxiety and surprise with the last exam were higher in genital warts group than for normal Pap smear and CIN groups

SECONDARY OUTCOMES:
economic burden of genital warts | January 2009 until December 2010
  Each genital wart episode lasted on average 132 ays, had 6 medical visits and costs US$ 139.

CONTACTS AND LOCATIONS:
Overall Officials: Monica G Almeida, MD, MS, Principal Investigator — BEMFAM Bem Estar Familiar no Brasil

IPD SHARING:
Plan to Share IPD: No